CLINICAL TRIAL: NCT05576389
Title: Neoadjuvant Fluzoparib Combined With Camrelizumab in Germline BRCA-mutated HER2-negative Breast Cancer: An Open-label, Single-arm, Multicenter Trial
Brief Title: Neoadjuvant Fluzoparib Combined With Camrelizumab in Germline BRCA-mutated HER2-negative Breast Cancer
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shu Wang, Chief Physician, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-035
Record Dates: First submitted 2022-09-13; First posted 2022-10-12 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Germline BRCA-mutated HER2-negative Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+Fluzoparib (Experimental)
  Interventions: Drug: Camrelizumab+Fluzoparib

INTERVENTIONS:
Drug: Camrelizumab+Fluzoparib — Fluzoparib：150mg was given orally twice daily Camrelizumab：200 mg IV drip on Day 1 of each cycle

SUMMARY:
This study is an open-label, single-arm, multicenter clinical study. 94 patients with germline BRCA-mutated HER2-negative early breast cancer are planned to be enrolled and treated with fluzoparib combined with camrelizumab to observe and evaluate the efficacy and safety of neoadjuvant fluzoparib combined with camrelizumab in the treatment of germline BRCA-mutated HER2-negative early breast cancer。

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 and ≤ 70 years of age with treatment-naïve breast cancer
* Histopathologically confirmed early or locally advanced HER2-negative invasive breast cancer as defined by the ASCO/CAP guidelines while meeting the following conditions:

HER2 negative: IHC 0/1 + or IHC2 + but ISH negative; Tumor stage: II-III; Primary tumor size: ≥ 1 cm Nodal Status: N0-3

* ECOG score 0 ~ 1;
* Centrally confirmed BRCA1 or BRCA2 germline mutation;
* At least one measurable lesion according to RECIST 1.1
* Eligible level of organ function

Exclusion Criteria:

* Patients with metastatic breast cancer or bilateral breast cancer;
* Patients with inflammatory breast cancer;
* Participated in other drug trials or received any anti-tumor therapy within 4 weeks before enrollment, including endocrine therapy, bisphosphonate therapy, immunotherapy, biological therapy or tumor embolization;
* Previously received PD-1/PD-L1 antibody, CTLA-4 antibody, or other therapies against PD-1/PD-L1 inhibitors;
* Previously received PARP inhibitors;
* Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS); active hepatitis or combined hepatitis B and C co-infection; autoimmune hepatitis;
* Confirmed history of heart failure or systolic dysfunction (LVEF < 50%); high risk uncontrolled cardiac arrhythmias, such as atrial tachycardia; angina requiring antianginal medication
* Female patients who are pregnant or lactating
* History of definite neurological or psychiatric disorders, including epilepsy or dementia
* Presence of interstitial lung disease, pneumonitis, or uncontrolled systemic disease (eg, diabetes mellitus, pulmonary fibrosis, acute pneumonitis, etc.)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
tpCR（ypT0/is ypN0） | 6 months
  total pathological complete response

CONTACTS AND LOCATIONS:
Overall Officials: Shu Wang, Dr., Principal Investigator — Breast Center, Peking University People's Hospital
Locations (1):
- Breast Cancer, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided